CLINICAL TRIAL: NCT02944305
Title: A New Prognostic Model Developed by Using Multi-predictive Tests for Prediction of Difficult Intubation in Adult Anesthetic Patients
Brief Title: A Predictive Model for Difficult Intubation
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Other Study IDs: HE581149
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Difficult Intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with difficult intubation: Group 1: Patient undergoing endotracheal intubation with difficult intubation Group 2: Patient undergoing endotracheal intubation without difficult intubation
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — Endotracheal intubation under direct laryngoscopy using McIntosh blade

SUMMARY:
Failure in airway management is one of the most common anesthesia-related morbidity and mortality. Each individual airway assessment has limitation to predict difficult intubation.

DETAILED DESCRIPTION:
Objective: To develop a scoring model from multiple airway assessment to predict difficult intubation.

Methods: This will be a retrospective analytic study. All airway assessment data from medical records of patients aged more than 18 years old underwent general anesthesia in Srinagarind hospital from January 2012 to December 2014 will be used to develop a new scoring prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing general anesthesia with endotracheal intubation

Exclusion Criteria:

* Incomplete airway assessment in medical record

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anesthesia with endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Difficult intubation | 5 minutes
  Laryngoscopic view: grade 1-2 = no difficult intubation; grade 3-4 = difficult intubation

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Result] Adnet F, Racine SX, Borron SW, Clemessy JL, Fournier JL, Lapostolle F, Cupa M. A survey of tracheal intubation difficulty in the operating room: a prospective observational study. Acta Anaesthesiol Scand. 2001 Mar;45(3):327-32. doi: 10.1034/j.1399-6576.2001.045003327.x. PMID 11207469
- [Result] Aktas S, Atalay YO, Tugrul M. Predictive value of bedside tests for difficult intubations. Eur Rev Med Pharmacol Sci. 2015;19(9):1595-9. PMID 26004598
- [Result] Iohom G, Ronayne M, Cunningham AJ. Prediction of difficult tracheal intubation. Eur J Anaesthesiol. 2003 Jan;20(1):31-6. doi: 10.1017/s0265021503000061. PMID 12553386
- [Result] Merah NA, Foulkes-Crabbe DJ, Kushimo OT, Ajayi PA. Prediction of difficult laryngoscopy in a population of Nigerian obstetric patients. West Afr J Med. 2004 Jan-Mar;23(1):38-41. doi: 10.4314/wajm.v23i1.28079. PMID 15171524